CLINICAL TRIAL: NCT01512537
Title: Comparison of UVB and Vitamin D Supplementation in Treatment of Vitamin D Deficiency
Brief Title: Alternative Treatments of Vitamin D Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Morten Bogh, Principal Investigator, Lund University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2009/687
Record Dates: First submitted 2011-12-22; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; UVB; Vitamin D supplementation
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- UVB (Active Comparator): UVB exposed group
  Interventions: Radiation: Narrowband UVB
- Oral vitamin D tablet (Active Comparator): Vitamin D supplementation
  Interventions: Dietary Supplement: Vitamin D and calcium

INTERVENTIONS:
Radiation: Narrowband UVB — UVB 3 times a week
  Other Names: NB-UVB
  Arms: UVB
Dietary Supplement: Vitamin D and calcium — 1 daily tablet of 1600 IU vitamin D3 and 1000 mg calcium
  Other Names: Vitamin D supplementation
  Arms: Oral vitamin D tablet

SUMMARY:
The purpose of the study is to compare the efficiency of UVB and vitamin D supplementation in treatment of vitamin D deficiency.

DETAILED DESCRIPTION:
Patients with vitamin D deficiency were recruited and randomized into two groups, one exposed to UVB and the other receiving oral treatment with vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin D deficiency (< 25 nmol/l)
* Age 15 or above

Exclusion Criteria:

* Travel south of 45 degrees latitude during the trial.
* Ongoing treatment with vitamin D supplementation.
* Intake of light sensitive medicine, such as tetracyclins.
* Skin light eruptions

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Vitamin D (nmol/l). | Week 0
  Vitamin D was measured in a bloodsample to determine baseline status.
Vitamin D (nmol/l) | Week 3
  Vitamin D was measured in a bloodsample to follow the change from baseline in vitamin D level at week 3.
Vitamin D | Week 6
  Vitamin D was measured in a bloodsample to follow the change from baseline in vitamin D level at week 6.

SECONDARY OUTCOMES:
Parathyroid hormone (pmol/l). | Week 0, 3 and 6.
  To investigate whether parathyrodiea hormone changes during the study.
Albumin (g/l). | Week 0, 3 and 6.
  To investigate whether albumin changes during the study.
Calcium (mmol/l) | Week 0, 3 and 6.
  To investigate whether calcium changes during the study.
Hemoglobin A 1c (percentage HbA1c of total hemoglobin). | Week 0, 3 and 6.
  To investigate whether HbA1c changes during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Åke Svensson, Assoc. Prof., MD, PhD, Study Chair — Department of Dermatology, Lund University, Malmoe
Locations (1):
- Department of Dermatology, Lund University Malmoe, Malmo, Sweden